CLINICAL TRIAL: NCT02661958
Title: A Phase 2, Randomized, Multicenter, Double-Blind, Active and Vehicle Controlled Parallel-group Study Evaluating the Efficacy, Safety, and Tolerability of Products S6G5T-3 and S6G5T-1 for the Treatment of Acne Vulgaris for 12 Weeks
Brief Title: Efficacy, Safety, and Tolerability of S6G5T-1 and S6G5T-3 for the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Collaborators: Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGT-65-02
Record Dates: First submitted 2016-01-11; First posted 2016-01-25 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- S6G5T-3 (Experimental): topical cream
  Interventions: Drug: S6G5T-3
- S6G5T-1 (Experimental): topical cream
  Interventions: Drug: S6G5T-1
- S6G5T-5 (Active Comparator): topical cream
  Interventions: Drug: S6G5T-5
- S6G5T-7 (Active Comparator): topical cream
  Interventions: Drug: S6G5T-7
- S6G5T-6 (Active Comparator): topical cream
  Interventions: Drug: S6G5T-6
- S6G5T-8 (Placebo Comparator): topical cream
  Interventions: Drug: S6G5T-8

INTERVENTIONS:
Drug: S6G5T-3 — once a day topical cream
  Arms: S6G5T-3
Drug: S6G5T-1 — once a day topical cream
  Arms: S6G5T-1
Drug: S6G5T-5 — once a day topical cream
  Arms: S6G5T-5
Drug: S6G5T-6 — once a day topical cream
  Arms: S6G5T-6
Drug: S6G5T-7 — once a day topical cream
  Arms: S6G5T-7
Drug: S6G5T-8 — once a day topical cream
  Arms: S6G5T-8

SUMMARY:
The purpose of this study is to evaluate the superiority in efficacy and assess safety and tolerability of the products S6G5T-3 and S6G5T-1 as compared to their respective active components or the vehicle for the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 9 years of age or older.
2. In good general health Based on medical records
3. Have a diagnosis of facial acne with >25 and <100 non-inflammatory lesions and >20 and <50 inflammatory lesions.
4. Have a score of "3" or "4" (Moderate or Severe) on the IGA scale.
5. Have two or fewer cysts or nodules (defined as an inflammatory lesion greater than or equal to 5 mm in diameter).
6. Sexually active women of child-bearing potential must use one of the following birth control options:

   One of these highly effective contraception methods:

   i. Intrauterine device (IUD); ii. Hormonal, for at least 3 months (Pills, injections, implants, transdermal patch, vaginal ring); iii. Tubal ligation; iv. Partner vasectomy,
7. OR A barrier form of contraception (listed below) i. Male or female condom; ii. Diaphragm with spermicides; iii. Cervical cap with spermicides; iv. Contraceptive sponge
8. Willingness and capacity for protocol compliance (for subjects under the age of consent, the parent/guardian must be willing and able to comply with study requirements).
9. Male subjects must be clean-shaven and agree to remain so for during the study visits.
10. Consent to participate, verified by signing an approved written Informed Consent Form and HIPAA; for subjects under the age of consent, both a signed assent form and a signed Informed Consent Form from the parent/guardian are required in accordance with local and federal regulations.

Exclusion Criteria:

1. More than two acne nodules or cysts (defined as an inflammatory lesion greater than or equal to 5 mm in diameter)
2. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc or severe acne requiring systemic treatment.
3. Underlying disease that requires the use of interfering topical or systemic therapy.
4. Other dermatological conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, atopic dermatitis, perioral dermatitis, or rosacea.
5. Beard, facial hair, or tattoo that may interfere with study assessments.
6. Use of tanning booths or tanning lamps within one week prior to Baseline and an unwillingness to refrain from use during the study.
7. Use of hormonal contraceptives, unless subject is on a stable dose for at least three months prior to enrollment.
8. Use of hormonal contraceptives solely for the control of acne.
9. Use of prohibited medications prior to the study and unwillingness to refrain from use during the study.
10. Known sensitivities to the study drug ingredients. Allergy to benzoyl peroxide, tretinoin, parabens and glycerin or other ingredients listed in the investigator brochure.
11. Clinically significant abnormal findings or conditions (other than acne), which might, in the opinion of the investigator, interfere with study evaluations or pose a risk to subject safety during the study.
12. Female subjects who are pregnant and/or nursing or planning to become pregnant during the course of the trial. Subjects who test positive for pregnancy after start of test treatment will be discontinued from test treatment but will be followed for safety purposes.
13. Participation in another investigational drug or device research study within 30 days of enrollment or five half-lives of the drug, whichever is longer.
14. Current or history of facial skin cancer.
15. Is an employee or family member of the study investigator or other study staff having direct involvement in the proposed study.
16. Is a family member of a study participant recruited and enrolled into the proposed study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2016-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) | week 12
  Proportion of subjects with an assessment of clear or almost clear with at least a 2-grade improvement in IGA at Week 12
Absolute change in lesion count (separately for inflammatory and non-inflammatory) | baseline and week 12
  Absolute change from Baseline in lesion count on the face at Week 12 (separately for inflammatory and non-inflammatory lesions)

SECONDARY OUTCOMES:
Percentage change from Baseline in lesion count on the face at Week 12 | Baseline and week 12
  Percentage change from Baseline in lesion count on the face at Week 12 (separately for inflammatory and non-inflammatory lesions)
assessments of IGA at each time point | baseline, week 4, 8
  Supportive efficacy variables are the assessments of IGA percentage change at each time point during the treatment period, namely at Weeks 4, and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Sheladia, M.S., Study Chair — Accelovance
Locations (34):
- United States (34):
  - Orange County Research Institute, Anaheim, California
  - Core Healthcare Group, Cerritos, California
  - eStudySite, Chula Vista, California
  - T. Joseph Raoof MD, Inc./Encino Research Center, Encino, California
  - Dermatology Research Associates, Los Angeles, California
  - eStudySite, Oceanside, California
  - Empire Clinical Research, Upland, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - MOORE Clinical Research, Inc, Brandon, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Oceane7 Clinical Research, Miami, Florida
  - RM Medical Research, LLC, Miami, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Dermatology Specialists Research, Louisville, Kentucky
  - DermResearch, PLLC, Louisville, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - MediSearch clinical Trials, Saint Joseph, Missouri
  - Quality Clinical Research Inc., Omaha, Nebraska
  - eStudySite, Las Vegas, Nevada
  - ActivMed Practices and Research, Inc., Portsmouth, New Hampshire
  - New York Clinical Trials, Manhattan, New York
  - Derm Research Center of New York, Inc, Stony Brook, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
  - Palmetto Clinical Trial Services, LLC @ Greenville Dermatology, Greenville, South Carolina
  - Discover Research, Inc., Bryan, Texas
  - West Houston Clinical Research Services LLC, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas